CLINICAL TRIAL: NCT01497002
Title: Randomized Phase III Study Comparing the OSHO Arm to the Standard Intergroup Arm.
Brief Title: Comparison of the OSHO Protocol to a Standard Arm Protocol of the German AML Intergroup in Patients With AML>60a
Acronym: AML2004
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSHO#069
Record Dates: First submitted 2011-12-21; First posted 2011-12-22 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2022-09

CONDITIONS: Acute Myeloid Leukaemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; TNK1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard arm (Active Comparator): standard treatment arm
  Interventions: Drug: Cytarabine
- OSHO - intensified consolidation (Experimental): Intermediate dose AraC
  Interventions: Drug: Cytarabine
- OSHO - allografting as consolidation (Experimental): allogeneic stem cell Transplantation versus no transplantation
  Interventions: Biological: human stem cells

INTERVENTIONS:
Drug: Cytarabine — Induction chemotherapy (1 or 2 courses): AraC 100 mg/m²/day i.v. 24h-infusion day 1-7 and Daunorubicin 60 mg/m² day 3+4+5. Consolidation chemotherapy (2 courses): AraC 1 g/m² i.v. 3h-infusion a 12h day 1+3+5.
  Other Names: AraC
  Arms: OSHO - intensified consolidation; standard arm
Biological: human stem cells — Induction chemotherapy (1 or 2 courses): AraC 1 g/m² i.v. 3h-infusion a 12h day 1+3+5+7, Mitoxantrone 10 mg/m² day 1-3 and Pegfilgrastim 6 mg s.c. day 10. Consolidation chemotherapy (1 course): AraC 500 mg/m² i.v. 1h-infusion a 12h day 1+3+5, Mitoxantrone 10 mg/m² day 1+2 and Pegfilgrastim 6 mg s.c. day 8. Allogeneic stem cell transplantation using reduced intensity conditioning: Fludarabine 30 mg/m² day -4 - -2, TBI 200 cGy day 0; GvHD prophylaxis: cyclosporine A and mofetil mycofenolate
  Arms: OSHO - allografting as consolidation

SUMMARY:
Improvement of the treatment-results in elderly patients with acute myeloid leukemia through intensification of consolidation chemotherapy and/or allografting as consolidative immunotherapy

DETAILED DESCRIPTION:
Measuring EFS depending on induction therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with age > 60 years and newly diagnosed acute myeloid leukaemia as defined by new WHO classification
* written informed consent

Exclusion Criteria:

* pretreatment of leukemia
* no informed consent
* simultaneous inclusion in other studies
* mental disability
* contraindication for intensive chemotherapy
* AML FAB M3
* contraindication for allogeneic stem cell transplantation
* restriction of following organ functions:
* creatinine-clearance < 50 ml/min
* cardiac ejection fraction < 40 %
* severe pulmonary restriction
* bilirubin > 2x ULN; SGOT and SGPT > 4x ULN
* uncontrolled hypertension
* severe uncontrolled metabolism disturbance
* Karnofsky-performance-score < 70%
* hepatitis C
* other malignancy
* age of unrelated donor >70 years and age of related donor >75 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1222 (Actual)
Dates: Start 2005-04 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Event free survival | after 5 years
  comparison of event free survival (OSHO arm versus Standard intergroup arm)

SECONDARY OUTCOMES:
OS | at 5 years
  Overall survival
LFS | at 5 years
  leukemia free survival

CONTACTS AND LOCATIONS:
Overall Officials: Dietger Niederwieser, Prof., Principal Investigator — University of Leipzig
Locations (1):
- University of Leipzig, Hematology, Leipzig, Germany

REFERENCES:
- See also: AML 2004 OSHO #069 (Elderly) — https://osho-studiengruppe.de/studie_069

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/02/NCT01497002/SAP_000.pdf